CLINICAL TRIAL: NCT04080219
Title: The Impact of Sleep-disordered Breathing on the Incidence of Postoperative Acute Kidney Injury in Patients Undergoing Valvular Heart Surgery: a Prospective Observational Study
Brief Title: The Impact of Sleep-disordered Breathing on the Incidence of Postoperative Acute Kidney Injury in Patients Undergoing Valvular Heart Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-1017
Record Dates: First submitted 2019-09-01; First posted 2019-09-06 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Valvular Heart Disease
Keywords: valvular heart surgery; cardiopulmonary bypass
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investigators measure the urinary NGAL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal: Patients with Oxygen desaturation index <5
- Sleep-disordered breathing: Patients with Oxygen desaturation index ≥5

SUMMARY:
Sleep-disordered breathing has a prevalence of 30~80% in patients with heart diseases. Various studies have revealed a correlation between the incidence and various diseases such as heart failure, hypertension, diabetes, and cerebral infarction. Postoperative acute kidney injury after heart surgery is one of the major complications with incidence with 40~50%, however, there has been no preventive method or treatment yet. Recently, several studies have been published that have shown a correlation between sleep-disordered breathing and renal impairment. In general, sleep-disordered breathing can be regulated easily with continues positive expiratory pressure, which means that early diagnosis and treatment of sleep-disordered breathing might help to reduce the incidence of postoperative acute kidney injury and improve patients' prognosis.

In this study, the investigators investigate the impact of sleep-disordered breathing (diagnosed by oxygen desaturation index ≥5) on the incidence of postoperative acute kidney injury in patients undergoing valvular heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient aged more than 20 years
2. Patients undergoing valvular heart surgery.

Exclusion Criteria:

1. Emergency
2. Simultaneous surgery with coronary artery bypass graft
3. Previous history of cerebrovascular accident
4. Previous history of sleep disordered breathing (diagnosis & treatment)
5. Previous history of tracheostomy
6. Previous history of surgical treatment of airway (ex: nasopharyngeal cancer)
7. Preoperative oxygen supplement therapy
8. Patients who have participated in other clinical studies that may affect prognosis
9. Patients who cannot read and agree to informed consent (ex: foreigners, cognitive dysfunction)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing valvular heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 414 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | Postoperative 7 days
  Postoperative acute kidney injury development defined by KDIGO criteria for postoperative 7 days.
  -KDIGO(Kidney Disease Improving Global Outcomes) is the global nonprofit organization developing and implementing evidence-based clinical practice guidelines in kidney disease.

SECONDARY OUTCOMES:
Urinary NGAL(Neutrophil gelatinase-associated lipocalin) by ELISA(enzyme-linked immunosorbent assay) | 15 minutes after anesthetic induction
  Urinary NGAL measurement by ELISA after anesthetic induction
Urinary NGAL(Neutrophil gelatinase-associated lipocalin) by ELISA(enzyme-linked immunosorbent assay) | Post-CPB 6hours
  Urinary NGAL measurement by ELISA after 6hours after cardiopulmonary bypass discontinuation
Urinary NGAL(Neutrophil gelatinase-associated lipocalin) by ELISA(enzyme-linked immunosorbent assay) | Post-CPB 24hours
  Urinary NGAL measurement by ELISA after 24hours after cardiopulmonary bypass discontinuation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No